CLINICAL TRIAL: NCT00976053
Title: Clinical Effectiveness of Pharmacologic Stress Radionuclide Myocardial Perfusion Imaging as a Guide to Management of Patients With Known CAD: Comparison of Single-Photon Emission Computed Tomography (SPECT) and Positron Emission Tomography (PET)
Brief Title: Effectiveness Study of Single Photon Emission Computed Tomography (SPECT) Versus Positron Emission Tomography (PET) Myocardial Perfusion Imaging
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aspire Foundation (Other)
Collaborators: Blue Cross Blue Shield (Other); Cardiovascular Imaging Technologies (Industry); Saint Luke's Cardiovascular Consultants (Other); Mid America Heart Institute (Other)
Responsible Party: Principal Investigator, Timothy M. Bateman, Prinicpal Investigator/Medical Director, Aspire Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-307
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Coronary Artery Disease
Keywords: Myocardial perfusion imaging; Single photon emission computed tomography; Positron emission tomography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SPECT myocardial perfusion imaging (Active Comparator)
  Interventions: Procedure: Myocardial perfusion imaging
- PET myocardial perfusion imaging (Active Comparator)
  Interventions: Procedure: Myocardial perfusion imaging

INTERVENTIONS:
Procedure: Myocardial perfusion imaging — Randomization assignment to one of SPECT or PET myocardial perfusion imaging

SUMMARY:
The purpose of this study is to compare pharmacologic stress myocardial perfusion PET with pharmacologic stress myocardial perfusion SPECT in a near-simultaneous, head-to-head comparison in the same patient. The investigators hypothesize that pharmacologic stress myocardial perfusion PET will prove superior to pharmacologic stress myocardial perfusion SPECT as a first-line diagnostic test for higher-risk patients with known coronary artery disease (CAD) who present with symptoms consistent with possible worsening of their CAD.

ELIGIBILITY:
Inclusion Criteria:

* History of coronary artery disease
* New or worsening symptoms
* Out-patients and in-hospital patients

Exclusion Criteria:

* Creatinine above 2.5 mg%
* PCI within prior 6 months
* Pregnant females
* Cardiomyopathy (LVEF below 40%)
* Significant valvular heart disease
* Body mass index greater than 38

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2009-06; Primary Completion 2013-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Diagnostic failure of SPECT vs PET | 60 days

SECONDARY OUTCOMES:
Composite of diagnostic or clinical failure | 12 months
Each of individual components of clinical failure | 12 months
Relative effect on quality of life | 3 months, 6 months
Relative direct and downstream costs | 3 months, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M Bateman, M.D., Principal Investigator — Aspire Foundation
Locations (1):
- Saint Luke's Cardiovascular Consultants, Kansas City, Missouri, United States

REFERENCES:
- [Derived] Patel KK, Al Badarin F, Chan PS, Spertus JA, Courter S, Kennedy KF, Case JA, McGhie AI, Heller GV, Bateman TM. Randomized Comparison of Clinical Effectiveness of Pharmacologic SPECT and PET MPI in Symptomatic CAD Patients. JACC Cardiovasc Imaging. 2019 Sep;12(9):1821-1831. doi: 10.1016/j.jcmg.2019.04.020. Epub 2019 Jul 17. PMID 31326480